CLINICAL TRIAL: NCT06071754
Title: Validation of the Performance of the Electrocardiogram (ECG) Function in the Masimo INVSENSOR00057
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Masimo Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: ECGV0001
Record Dates: First submitted 2023-09-18; First posted 2023-10-06 (Actual); Results first posted 2025-06-12 (Actual); Last update posted 2025-10-31 (Actual); Status verified 2025-10

CONDITIONS: Healthy; Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- INVSENSOR00057 (Experimental): All subjects are enrolled into this arm and will have ECG measurements obtained
  Interventions: Device: Masimo INVSENSOR00057

INTERVENTIONS:
Device: Masimo INVSENSOR00057 — Masimo INVSENSOR00057 will be used to collect electrocardiogram measurements.

SUMMARY:
The objective of this study is to validate the performance of the electrocardiogram (ECG) function of the Masimo INVSENSOR00057 against contemporaneous measurements

ELIGIBILITY:
Inclusion Criteria:

* Subject is 22 years of age or older
* Subject is comfortable to read and communicate in English*
* Subject belongs to one of two groups:
* Subjects without any prior arrhythmia diagnosis presenting in normal sinus rhythm (Group1)
* Subjects with history of paroxysmal or persistent atrial fibrillation presenting in atrial fibrillation (Group 2) *This is to ensure the subject can provide informed consent (as Masimo INVSENSOR00057 ECG study materials are currently available in English only) and can comply with study procedures.

Exclusion Criteria:

* Subjects who are physically unable to wear a wristwatch
* Subjects whose skin is not intact (e.g., has open wounds, has inflamed tattoos or piercings, has visible healing wounds) in or at the vicinity of the device placement site.
* Subjects with an implantable defibrillator or cardiac pacing device.
* Subjects with a skin condition which would preclude proper ECG electrode placement..
* Subjects with known allergic reactions to adhesive tapes or ECG gel.
* Subjects previously diagnosed with non-atrial fibrillation cardiac arrhythmia.
* Subjects not suitable for the investigation at the discretion of the investigator or the clinical team

Min Age: 22 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 365 (Actual)
Dates: Start 2023-09-01 (Actual); Primary Completion 2024-04-30 (Actual); Study Completion 2024-04-30 (Actual)

CONTACTS AND LOCATIONS:
Locations (4):
- United States (4):
  - Masimo Clinical Lab, Irvine, California
  - PCA Cardiology, Laguna Hills, California
  - Cone Health, Greensboro, North Carolina
  - Medication Management, Greensboro, North Carolina

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | INVSENSOR00057
Started | 365
Completed | 356
Not Completed | 9
Not completed — Device rhythm classifications not obtained from subjects due to protocol not being completed | 9

BASELINE CHARACTERISTICS:
Arm/Group | INVSENSOR00057
Number analyzed (Participants) | 365
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 199
  >=65 years | 166
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 140
  Male | 225
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Hispanic, Latino or Spanish | 55
  Non-Hispanic, Latino or Spanish | 259
  Not Reported | 51
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 58
  Black or African American | 26
  Native Hawaiian or Other Pacific Islander | 2
  White | 209
  Other | 31
  Not Reported | 39

OUTCOME MEASURES:

1. Primary Outcome: Validation of the Performance of the Electrocardiogram (ECG) Function in the Masimo INVSENSOR00057
Description: Single Lead ECG, similar to lead I, intended to be used for Heart Rate measurement and AFib detection
Time Frame: Approximately 30 minutes
Population: Masimo W1 rhythm classifications were not obtained from 9 subjects (3 from the NSR group, 6 from AFib group) due to the subject not completing the protocol.
Measure: Number; unit: percent
Arm/Group | INVSENSOR00057
Number analyzed (Participants) | 356
percent
  Sensitivity | 99.3
  Specificity | 100.0

ADVERSE EVENTS:
Time Frame: 30 minutes
Description: Definitions do not differ
Arm/Group | INVSENSOR00057
All-Cause Mortality (participants affected / at risk) | 0/365
Serious Adverse Events (participants affected / at risk) | 0/365
Other Adverse Events (participants affected / at risk) | 0/365

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-04-16): https://cdn.clinicaltrials.gov/large-docs/54/NCT06071754/Prot_SAP_000.pdf